CLINICAL TRIAL: NCT04376541
Title: Fast Tracking Impact on Fentanyl Consumption and Parents Satisfaction in Non Complex Cardiac Surgery
Brief Title: Fast Tracking Impact on Fentanyl Consumption and Parents Satisfaction
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Gamal Adel Adelhameed, lecturer of anesthesia and intensive care and pain management, Ain Shams University
Other Study IDs: s 43
Record Dates: First submitted 2020-04-28; First posted 2020-05-06 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-05

CONDITIONS: Fentanyl Adverse Reaction; Caudal Anesthesia
Keywords: fast track; congenital cardiac surgery; caudal; fentanyl
MeSH Terms: interventions — Fentanyl

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- early extubation: the patients extubated in O.R or within 2 hours in the ICU
  Interventions: Drug: Fentanyl
- late extubation: the patients extubated after 2 hours from O.R
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Fentanyl — amount of fentanyl used in both groups

SUMMARY:
The investigators are measuring fentanyl consumption in micrograms used during anesthesia for patients on fast track congenital cardiac surgeries

DETAILED DESCRIPTION:
The investigators are measuring fentanyl consumed for both fast track and conventional corrective cardiac surgeries and also parents Parental Perceptions satisfaction with early child communication in ICU and impact of caudal anesthesia on extubation time our 2ry outcomes are the hospital and ICU length of stay

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with congenital cardiac anomaly for surgical correction.
* age limit: child 3months of age to 18 years

Exclusion Criteria:

patients with any o the following:

* emergency surgeries
* redo surgeries
* complex surgeries
* patients weight less than 3kg

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: patients diagnosed with congenital cardiac anomaly for surgical correction from 3months to 18 years of age
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
fentanyl consumption | during the procedure (corrective surgery)
  amount of fentanyl used in microgram
parents satisfaction: questionnare | after discharge from the ICU up to 1 week
  questionnare for parents satisfaction by early child communication

SECONDARY OUTCOMES:
intensive care length of stay | after departure from operation room until ward discharge up to 3 weeks
  number of days in ICU
hospital length of stay | from admission until home discharge up to 4 weeks
  total number of days spent in hospital

IPD SHARING:
Plan to Share IPD: Undecided
IPD Will be shared upon request